CLINICAL TRIAL: NCT05040308
Title: Implementation Science Research on PrEP Delivery and Costing Within Harm Reduction Services for People Who Use Drugs in Uganda
Brief Title: Uganda PrEP and Harm Reduction Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Makerere University (Other)
Responsible Party: Principal Investigator, Renee Heffron, Associate Professor, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00012972; R01DA051796 (NIH)
Record Dates: First submitted 2021-05-20; First posted 2021-09-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-04

CONDITIONS: HIV-1-infection
Keywords: pre-exposure prophylaxis; substance use disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants in PrEP and MAT programs (Active Comparator): Integrated PrEP and MAT program
  Interventions: Other: Integrating PrEP delivery
- Participants in PrEP and NSP programs (Active Comparator): Integrated PrEP and NSP program
  Interventions: Other: Integrating PrEP delivery

INTERVENTIONS:
Other: Integrating PrEP delivery — Integration of PrEP delivery services in NSP and MAT programs

SUMMARY:
This is an evaluation of programs to integrate PrEP into existing services for PWUD. PrEP will be delivered according to Uganda national guidelines and data from national monitoring and evaluation forms will be leveraged to address key outcomes. Additionally, research components will be implemented to support greater understanding of PrEP use and experiences of participants engaged with the PrEP programs.

DETAILED DESCRIPTION:
The first facility-based medication-assisted treatment (MAT) program (with methadone) in Kampala launched in 2020, providing opportunity to integrate pre-exposure prophylaxis(PrEP) as part of a comprehensive HIV prevention package. Additionally, a community-based needle and syringe exchange program (NSP) provides opportunity to integrate PrEP and meet priorities of PWID while building rapport between providers and end-users. With two different service models - integrating PrEP into facility-based MAT and community-based NSP - there is a great opportunity to optimize the integration of PrEP and other HIV prevention services for PWUD. By integrating PrEP into two existing programs (MAT and NSP), this study will determine uptake and persistence of PrEP use and leverage these programs to conduct costing research and budget impact analysis.

ELIGIBILITY:
Inclusion Criteria:

* Accessing services from any of the programs implementing the integrated PrEP program described in this protocol
* Able and willing to provide informed consent
* Age ≥15 years

Exclusion Criteria:

* Any clinical or chronic medical condition that in the opinion of the investigator would make the participant unsuitable for the study or unable to independently provide informed consent.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of PrEP uptake | 12 months after enrollment
  PrEP uptake will be measured through PrEP bottle inventory (bottles dispensed) in people who access NSP versus MAT.
PrEP retention | 12 months after enrollment
  PrEP retention will be measured through study visit attendance among those who access NSP versus MAT.
PrEP adherence | 12 months after enrollment
  PrEP adherence will be measured objectively through plasma tenofovir in people who access NSP versus MAT.

SECONDARY OUTCOMES:
To measure the impact of knowledge gained from training peers of PWUD on PrEP. | Baseline (pre-training), immediately after training, and 3 months post training
  The clinic staff will train up to 50 health care providers of PWUD on PrEP service delivery using the national curriculum on PrEP services delivery. We will administer a quantitative assessment of PrEP knowledge and experiences with service provision at three time points: 1. Before the training (Baseline survey), 2. immediately after training (Post training survey), and 3. ~3 months post training (Exit survey).
To conduct a budget impact analysis for integrating PrEP into MAT and NSP programs. | 12 months post study enrollment
  The clinic staff will conduct micro costing c using activity-based approaches for costs incurred (clinic wide trainings, recruitment, service delivery, lab monitoring, PrEP support, and provision of PrEP) and costs averted (health costs saved by averting incident HIV infections). Cost data will also be collected from the study budget, public health clinic budgets, published government reports, and the health economics literature. Time and motion studies will be conducted by observing visits of people who are accessing services, and staff time spent on counseling, clinical procedures, and delivering PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Heffron, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Diseases Institute, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No